CLINICAL TRIAL: NCT04001673
Title: Impact of a Pharmacist's Intervention on Knowledge and Adherence to Biologic Disease-modifying Drugs in Patients With Spondyloarthritis: a Randomised Controlled Trial.
Brief Title: Pharmaceutical Intervention and Adherence to bDMARDs in Spondyloarthritis.
Acronym: SPADHESION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Ornella Conort (Other)
Responsible Party: Sponsor-Investigator, Dr Ornella Conort, Pharmacist, Hôpital Cochin
Organization: Hôpital Cochin (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-A01897-44
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Spondyloarthritis; Treatment Adherence
Keywords: treatment knowledge
MeSH Terms: conditions — Spondylarthritis; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist's intervention (Active Comparator): Evaluation of knowledge and adherence of patients treated by bDMARDs before and after the intervention of a pharmacist that will give information concerning bDMARDs management.
  Interventions: Behavioral: Pharmacist's intervention
- Control (No Intervention): Evaluation of knowledge and adherence of patients treated by bDMARDs who did not receive pharmacist's intervention.

INTERVENTIONS:
Behavioral: Pharmacist's intervention — Information about bDMARDs management.
  Arms: Pharmacist's intervention

SUMMARY:
There is a lack of knowledge among patients concerning their treatment with bDMARDs, which could lead to low adherence.

The objective of this study is to assess the impact of a pharmacist's intervention on the adherence to bDMARDs in patients with Spondyloarthritis.

DETAILED DESCRIPTION:
This is an interventional, controlled, open-label and monocentric study. 80 patients are planned to be included.

After written informed consent will be obtained, the patients will be randomized in two arms:

* Intervention arm: intervention of a pharmacist who will explain bDMARDs management.
* Control arm, without intervention.

Two primary end-points are defined:

1. the changes from baseline to M6 in the patients' knowledge score about subcutaneous bDMARD management
2. the changes from baseline to M6 in Medication Possession Ratio (MPR)

As secondary end-points, the changes in disease activity and patients' satisfaction regarding the pharmacists' intervention are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients from Rheumatology Department at Cochin Hospital
* Diagnosis of Spondyloarthritis
* Under treatment with subcutaneous bDMARDs for at least 6 months
* Disease activity stable for at least 6 months
* No treatment modification 3 months before or after inclusion in the study
* Informed consent signed and dated
* Older than 18 years
* Patients who speak french

Exclusion Criteria:

* Patients who have had a change in the treatment of SpA during the 3 months prior or after the inclusion
* History of psychological problems
* Patients who need other persons to manage their treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Improvement in bDMARDS adherence at 6 months in patients who received a pharmaceutical intervention. | 6 months of follow-up
  MPR score comparison between the two arms after 6 month of follow up. MPR represents the number of subcutaneous bDMARDs supplied by a pharmacy divided by the number of theorical subcutaneous bDMARDs that the patient should have taken within the observation period (e.g. during the 4 months preceeding the baseline or the M6 visit), expressed in percentage.
Improvement in knowledge about bDMARDs management. | 6 months of follow-up
  Knowledge level comparison (well-known, not known, partially known) evaluated by self-questionnaire between the two arms after 6 months of follow-up.

SECONDARY OUTCOMES:
Changes in disease activity | 6 months of follow-up
  BASDAI score comparison between the two arms after 6 month of follow up.
Satisfaction of patients after receiving pharmacist's intervention | 6 months of follow-up
  Answer comparison to the 4-Likert self-questionnaire between the two arms after 6 months of follow-up. The Likert Scale is a four point scale, from not at all satisfied to completely satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Cochin, Paris, Ille de France, France

IPD SHARING:
Plan to Share IPD: No